CLINICAL TRIAL: NCT05821582
Title: Study SBX-01-101: A Stool Collection Study in Colorectal Cancer (CRC) Patients Treated With Irinotecan-Based Regimens
Status: Withdrawn | Type: Observational
Why Stopped: Insufficient recruitment population.
Sponsor: Sanguine Biosciences (Industry)
Responsible Party: Sponsor
Other Study IDs: SAN-09391
Record Dates: First submitted 2023-03-21; First posted 2023-04-20 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Stool Collection and Survey Completion — Participants will have 2 scheduled at-home stool self-collections at the time points specified in section 4.0 and complete a questionnaire by telephone contact. The biospecimens collected from participants on this study are stool samples.

SUMMARY:
The primary objective of the study is to determine whether there is a correlation between the intestinal side effects of chemotherapy treatment and the expression/activity profiles of glucuronidase enzymes in the stool microbiome of the target patient population.

DETAILED DESCRIPTION:
STUDY DESIGN:

* This protocol is a single-center, single-cohort, bioresearch study enrolling up to 8 participants. The cohort is as follows:
* Cohort 1: Colorectal Cancer: (n=8)
* The study will enroll participants per the eligibility criteria.
* Participants will have 2 scheduled at-home stool self-collections at the time points specified in section 4.0 and complete a questionnaire by telephone contact (see section 11.0 for details). The biospecimens collected from participants on this study are stool samples.
* Confirmation of eligibility and medical record review by a member of the study staff will be completed for participants of the disease cohort before they are considered fully enrolled.

ELIGIBILITY:
Cohort 1: Colorectal Cancer

Inclusion:

1. The participant is willing and able to provide written informed consent
2. The participant is willing and able to provide appropriate photo identification
3. Participants aged 18 to 85, Inclusive
4. Participants have been diagnosed with Active Colorectal Cancer (CRC)
5. Subjects currently taking irinotecan

Exclusion:

1. Participants who are pregnant or are nursing
2. Participants with a known history of HIV, hepatitis, or other infectious diseases
3. Participants who have taken an investigational product in the last 30 days
4. Participants who have experienced excess blood loss, including blood donation, defined as 250 mL in the last month or 500 mL in the previous two months
5. Subjects who are currently in remission for CRC.

   * Preference (not required for enrollment into study): Exclude subjects currently taking antibiotics*

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with active colorectal cancer
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-10-05 (Actual); Study Completion 2023-10-05 (Actual)

PRIMARY OUTCOMES:
Primary Objective- Intestinal side effects of chemotherapy | 8 months
  The primary objective of the study is to collect stool samples to provide to the sponsor so the sponsor can assess whether there is a correlation between the intestinal side effects of chemotherapy treatment and the expression/activity profiles of glucuronidase enzymes in the stool microbiome of the target patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew C Frisina, M.S., Study Director — Sanguine Biosciences
Locations (1):
- Sanguine Biosciences, Inc., Woburn, Massachusetts, United States